CLINICAL TRIAL: NCT06240494
Title: Predictive Factors Associated With Successful Response to Ultrasound-guided Maxillary and Mandibular Nerve Radiofrequency Treatment for Trigeminal Neuralgia
Brief Title: Predictive Factors in Maxillary and Mandibular Nerve Radiofrequency Treatment for Trigeminal Neuralgia
Status: Completed | Type: Observational
Sponsor: Diskapi Teaching and Research Hospital (Other)
Responsible Party: Principal Investigator, Damla Yürük, Medical doctor, Diskapi Teaching and Research Hospital
Other Study IDs: Maxillary and mandibular RF
Record Dates: First submitted 2024-01-26; First posted 2024-02-05 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Trigeminal Neuralgia
Keywords: mandibular nerve; maxillary nerve; pulsed radiofrequency; ultrasound; analgesia
MeSH Terms: conditions — Trigeminal Neuralgia; Agnosia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Maxillary nerve and mandibular nerve pulsed radiofrequency — For maxillary nerve pulsed radiofrequency, the lineer transducer is placed distal and parallel to the zygomatic arch, bridging the coronoid and condylar processes and a 22 gauge 6 mm RF cannula was inserted into the target area. With sensory stimulation, patients experienced a distinct sensation in upper jaw, teeth, and palate. Then, PRF treatment was performed at 42 °C for 240 seconds.
  For mandibular nerve pulsed radiofrequency, the transducer was placed distally and parallel to the zygomatic arch, bridging the coronoid and condylar processes. The pterygopalatine fossa was visualized and the needle was inserted to target area. With sensory stimulation, patients experienced a distinct sensation in the lower jaw and teeth. With motor stimulation, a throwing movement of the jaw was observed with contraction of the masseter and temporal muscles. PRF treatment was performed at 42 °C for 240 s.

SUMMARY:
Trigeminal neuralgia is one of the most common craniofacial neuralgias and one of the most severe types of facial pain, typically limited to the distribution of the trigeminal nerve. The first-line treatment for trigeminal neuralgia is medical therapy and primarily antiepileptic drugs. Various interventional and surgical methods can be used in patients who do not respond to medical treatment or who cannot tolerate side effects. Pulsed radiofrequency treatment of maxillary and mandibular nerves may provide longer-lasting pain relief in trigeminal neuralgia.This study aimed to investigate the clinical and demographic characteristics affecting treatment success in patients who underwent ultrasound-guided pulsed radiofrequency of the maxillary and/or mandibular nerves for trigeminal neuralgia.

DETAILED DESCRIPTION:
Pulsed radiofrequency treatment applied to the maxillary and mandibular nerves, which are the peripheral branches of the trigeminal nerve, is frequently used in patients with trigeminal neuralgia who do not adequately respond to medical treatment.

Pain intensity was evaluated at baseline and 3 months after US-guided maxillary and/or mandibular nerve PRF treatment using NRS (numerical rating scale). The primary outcome measure was percent reduction in pain, with 50% pain relief lasting at least 3 months was defined as a positive categorical outcome.

In addition, demographic data such as age (years), gender, duration of pain (months), etiology (idiopathic or secondary), MRI findings (normal findings or abnormal findings due to conditions such as vascular compression and demyelinating plaque), pain side (unilateral or bilateral), and history of Gasser ganglion RF ablation were obtained from patient data. NRS scores before and 3 months after PRF were collected from the patient data and recorded. Pre-procedural cranial MRI and MR cisternography reports were accessed from patient records, and any abnormalities were recorded. We retrospectively analyzed the patient's electronic medical history records and the archive system containing the imaging results to obtain the variables.

The main aim of this study was to determine the clinical and demographic variables associated with treatment outcomes in patients with TN who underwent PRF of the maxillary and mandibular nerves. The secondary aim of this study was to determine the incidence of procedure-related adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of trigeminal neuralgia according to the IHS 3-beta criteria
* No response to conservative treatment for > 3 months
* Magnetic resonance imaging within 1 year prior to injection
* Access to clinical data

Exclusion Criteria:

* Inadequate medical records with missing numerical rating scale (NRS) scores and MRI images
* Patients lost to follow-up within three months after the procedure
* History of surgery or gamma-knife radiosurgery for trigeminal neuralgia
* History of malignancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female patients who underwent maxillary and/or mandibular nerve pulsed radiofrequency for trigeminal neuralgia
Sampling Method: Non-Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-02 (Actual)

PRIMARY OUTCOMES:
VAS | Change from Baseline NRS at 3 months
  Visual analogue scales (VAS) are psychometric measuring instruments designed to document the characteristics of disease-related symptom severity in individual patients and use this to achieve a rapid (statistically measurable and reproducible) classification of symptom severity and disease control.

CONTACTS AND LOCATIONS:
Overall Officials: Ömer Taylan Akkaya, MD, Principal Investigator — Diskapi Teaching and Research Hospital; Ezgi Can, MD, Study Director — Diskapi Teaching and Research Hospital
Locations (1):
- Ankara Etlik City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided